CLINICAL TRIAL: NCT02518490
Title: A Contralateral Dispensing Clinical Trial of Study Test Sapphire Lens Against Enfilcon A Silicone Hydrogel Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV-15-46
Record Dates: First submitted 2015-08-04; First posted 2015-08-07 (Estimated); Results first posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Sapphire lens (Experimental): Each subject will be randomized to wear the test lens on one eye and control lens on one eye.
  Interventions: Device: Sapphire Lens
- enfilcon A (Active Comparator): Each subject will be randomized to wear the test lens on one eye and control lens on one eye.
  Interventions: Device: enfilcon A

INTERVENTIONS:
Device: Sapphire Lens — Each subject will be randomized to wear the test lens on one eye and control lens on one eye.
  Arms: Sapphire lens
Device: enfilcon A — Each subject will be randomized to wear the test lens on one eye and control lens on one eye.
  Arms: enfilcon A

SUMMARY:
This was be a randomized, contralateral, double-masked, dispensing study comparing the Study test lens against the control lens over one month of lens wear.

The study results were not used for design validation of test lens.

DETAILED DESCRIPTION:
Subjects were randomized to wear the test lens in one eye and control lens in the other eye. Both test and control lenses were used in a daily wear modality for one month.

The study results were not used for design validation of test lens.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will only be eligible for the study if:

  1. Is at least 18 years of age for the USA and has full legal capacity to volunteer;
  2. Has read and signed an information consent letter;
  3. Is willing and able to follow instructions and maintain the appointment schedule;
  4. Is an adapted soft contact lens wearer;
  5. Requires spectacle lens powers between -0.50 to -6.50 diopters sphere;
  6. Has no more than 0.75 diopters of refractive astigmatism;
  7. Willing to wear contact lens in both eyes;
  8. Has manifest refraction visual acuities (VA) equal to or better than logMAR equivalent of 20/25 in each eye;
  9. To be eligible for lens dispensing, the subject must have VA of logMAR equivalent of 20/30 or better in each eye with the study lenses and the investigator must judge the fit as acceptable.

     Exclusion Criteria:
* Subjects will not be eligible to take part in the study if:

  1. Is participating in any concurrent clinical or research study;
  2. Has any known active* ocular disease and/or infection;
  3. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
  4. Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
  5. Has known sensitivity to the diagnostic pharmaceuticals to be used in the study;
  6. Is pregnant, lactating or planning a pregnancy at the time of enrolment (by verbal confirmation at the screening visit);
  7. Is aphakic;
  8. Has undergone refractive error surgery; * For the purposes of this study, active ocular disease is defined as infection or inflammation which requires therapeutic treatment. Mild (i.e. not considered clinically relevant) lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining and dry eye are not considered active ocular disease. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-08; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meng Lin, Principal Investigator — Clinical Research Center, University of California, Berkeley
Locations (1):
- Clinical Research Center, University of California, Berkeley, Berkeley, California, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Groups:
- Sapphire Lenses: Each subject will be randomized to wear the test lens in one eye and control lens in the other eye. Both test and control lenses will be used in a daily wear modality for one month.
  Sapphire Lens: Contact Lenses
- Enfilcon A: Each subject will be randomized to wear the test lens in one eye and control lens in the other eye. Both test and control lenses will be used in a daily wear modality for one month.
  enfilcon A: Contact lenses
Period: Overall Study
Arm/Group | Sapphire Lenses | Enfilcon A
Started | 18; 18 Eyes | 18; 18 Eyes
Completed | 17; 17 Eyes | 17; 17 Eyes
Not Completed | 1; 1 Eyes | 1; 1 Eyes
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: 18 subjects were fit with study lenses and one subject discontinued at the dispensing visit due to dissatisfaction with both study lenses. Baseline demographic information is gathered for 17 subjects.
Groups:
- Overall Study: Subjects were randomized to wear test lens in one eye and control lens in other eye for a one month period.
Arm/Group | Overall Study
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Subjective Ratings for Comfort After Lens Insertion
Description: Subjective ratings for comfort on a scale (0-100) assessed : 0= Cannot be worn, causes pain, 20=Frequently irritating, 40= Occasionally irritating, 60= Occasionally noticable but not irritating, 80= rarely noticeable, 100= cannot be felt ever
Time Frame: Baseline (5 minutes post lens dispensing)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Sapphire Lenses | Enfilcon A
Number analyzed (Participants) | 17 | 17
Number analyzed (Eyes) | 17 | 17
units on a scale | 91 (11) | 93 (12)

2. Primary Outcome: Subjective Ratings for Comfort After Lens Insertion
Description: as for outcome 1
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Sapphire Lenses | Enfilcon A
Number analyzed (Participants) | 17 | 17
Number analyzed (Eyes) | 17 | 17
units on a scale | 88 (11) | 87 (15)

3. Primary Outcome: Percentage of Participants With a Lens Preference Based on Subjective Comfort
Description: Percentage of Participants with a Lens Preference Based on Subjective Comfort. Preferred Sapphire, Preferred Enfilcon A, No preference
Time Frame: Baseline (5 minutes post lens dispensing)
Measure: Number; unit: percentage of participants
Groups:
- Overall Study: Subjects were randomized to wear test lens in one eye and control lens in other eye for a one month period.
  Sapphire Test lens: Contact lens Enfilcon A: contact lens
Arm/Group | Overall Study
Number analyzed (Participants) | 17
percentage of participants
  Sapphire | 20
  No preference | 30
  enfilcon A | 50

4. Primary Outcome: Percentage of Participants With a Lens Preference Based on Subjective Comfort
Description: as for outcome 3
Time Frame: 4 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study
Number analyzed (Participants) | 17
percentage of participants
  Sapphire | 10
  No preference | 65
  enfilcon A | 25

5. Primary Outcome: Lens Wettability
Description: Lens wettability was assessed on a Grading scale (0-4, 0.25 steps) (0=excellent; 4=severely reduced)
Time Frame: Baseline (5 minutes post lens dispensing)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Sapphire Lenses | Enfilcon A
Number analyzed (Participants) | 17 | 17
Number analyzed (Eyes) | 17 | 17
units on a scale | 3.4 (0.4) | 3.4 (0.3)

6. Primary Outcome: Lens Wettability
Description: Lens wettability was assessed on a Grading scale (0-4, 0.25 steps) (0=excellent; 4=severely reduced)
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Sapphire Lenses | Enfilcon A
Number analyzed (Participants) | 17 | 17
Number analyzed (Eyes) | 17 | 17
units on a scale | 3.5 (0.4) | 3.6 (0.3)

7. Primary Outcome: Lens Surface Deposition
Description: Lens Surface Deposit was assessed on a scale of 0-4 (0-4, 0.25 steps)(0- Clean , no deposits, 1- 5 or less small deposits (<0.1mm), 2- >5 deposits of <0.1mm size or film covering 25-50% of surface, 3 - Deposits of between 0.1 and 0.5amm or film covering 50-75% of surface, 4- Deposits of 0.5mm or larger or film covering more than 75% of surface)
Time Frame: Baseline (5 minutes post lens dispensing)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Sapphire Lenses | Enfilcon A
Number analyzed (Participants) | 17 | 17
Number analyzed (Eyes) | 17 | 17
units on a scale | 0.06 (0.17) | 0.03 (0.12)

8. Primary Outcome: Lens Surface Deposition
Description: as for outcome 7
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Sapphire Lenses | Enfilcon A
Number analyzed (Participants) | 17 | 17
Number analyzed (Eyes) | 17 | 17
units on a scale | 0.21 (0.50) | 0.10 (0.27)

ADVERSE EVENTS:
Time Frame: From dispense up to 4 weeks on the study lenses.
Arm/Group | Sapphire Lenses | Enfilcon A
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No